CLINICAL TRIAL: NCT05308823
Title: Outcome of Cerebral Venous Sinuses Stenting on Idiopathic Intracranial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alwathekbellah Ihab Ahmed Elsayed, Doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000046
Record Dates: First submitted 2022-02-11; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: Idiopathic Intracranial Hypertension stenting
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Stents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): The paients in this group will receive traditional treatment of IIH for 3 months.
- Group 2 (Experimental): The patients in this group will receive traditional treatment of IIH for 3 months in addition to venus sinus stent.
  Interventions: Procedure: Stent

INTERVENTIONS:
Procedure: Stent — The patients in this group will receive traditional treatment of IIH for 3 months in addition to venus sinus stent
  Other Names: Venous sinus stenting
  Arms: Group 2

SUMMARY:
The aim of the work is to asses the positive effect of stenotic sinus segment stenting on idiopathic intracranial hypertension with headache and papilloedema.

DETAILED DESCRIPTION:
Participants The study will include group of patients with an established diagnosis of idiopathic intracranial hypertenton meeting our inclusion criteria and will admitted to Al-Azher Univerity Hospitals (Al-Hussien and Bab El-Shaeria) after informed consent from them. The recruitment will take place after approval from the Ethics Committee and the University Council.

* They are selected according to The modified Dandy Criteria to Diagnose IIH:

  1. Grade II paplledema .
  2. normal neurological examination except for six nerve palsy.
  3. neuroimaging criteria of normal brain parenchyma without evidence of hydrocephalus, mass or structural lesion and no abnormal meningeal enhancement on MRI.
  4. normal CSF composition.
  5. elevated lumbar puncture opening pressure, defined as greater than or equal to 250 mmH2O in adults (7).
* Exclusion criteria included:

  1. Age less than orequal to 18 years.
  2. creatinine .1.5 mg/dL.
  3. severe allergic reaction to iodine contrast.
  4. contraindication to general anesthesia, use of aspirin, clopidogrel or anticoagulants, thrombophilic disorder or anticardiolipin syndrome.
  5. dural arteriovenous fistula or other arteriovenous lesion affecting cortical venous flow.
  6. pregnancy.
  7. Blood pressure must be measured to exclude malignant hypertension, as defined as a diastolic blood pressure greater than or equal to 120 mm Hg or systolic blood pressure greater than or equal to 180 mm Hg(17).

ELIGIBILITY:
Inclusion Criteria:

* 1. Grade II paplledema . 2. normal neurological examination except for six nerve palsy. 3. neuroimaging criteria of normal brain parenchyma without evidence of hydrocephalus, mass or structural lesion and no abnormal meningeal enhancement on MRI. 4. normal CSF composition. 5. elevated lumbar puncture opening pressure, defined as greater than or equal to 250 mmH2O in adults

Exclusion Criteria:

* 1. Age less than to 18 years. 2. creatinine .1.5 mg/dL. 3. severe allergic reaction to iodine contrast. 4.contraindication to general anesthesia, use of aspirin, clopidogrel or anticoagulants, thrombophilic disorder or anticardiolipin syndrome. 5. dural arteriovenous fistula or other arteriovenous lesion affecting cortical venous flow. 6. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-09-05 (Estimated)

PRIMARY OUTCOMES:
Change in papillodema | 3 months after intervention
  Frisen scale in grading of papilledema evaluation
Improvement of headache | 3 months after intervention
  Headache Impact Test (HIT-6) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ahmed Zaki, Ass. Prof, Study Director — Al-Azher Univerity Hospitals (Al-Hussien and Bab El-Shaeria)
Locations (1):
- Al-Azher Univerity Hospitals (Al-Hussien and Bab El-Shaeria), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
All selected patients will be assessed after 3 months for headache and papilledema by (HIT-6) questionnaire in headache evaluation and Frisen scale in grading of papilledema evaluation in addition to MRV.